CLINICAL TRIAL: NCT05472272
Title: Effect of Low-Calorie Diets on Remission of Type 2 Diabetes: A Feasibility Study
Brief Title: Low-Calorie Diets on Type 2 Diabetes Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Feng Tao, Director, Shanghai Municipal Hospital of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHMHTCM DM
Record Dates: First submitted 2022-07-09; First posted 2022-07-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Overweight
Keywords: Type 2 diabetes; Diabetes mellitus; Weight loss; Diet; Lifestyle intervention; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Diabetes Mellitus; Weight Loss | interventions — Food, Formulated

STUDY DESIGN:
Intervention Model Description: This is a non-randomized parallel study without a control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula Diet (Experimental): Participants will receive a low-calorie formula diet product.
  Interventions: Other: Formula diet
- Food-Based Diet (Experimental): Participants will receive a low-calorie food-based diet created by dietitians.
  Interventions: Other: Food-based diet

INTERVENTIONS:
Other: Formula diet — Participants will receive a low-calorie (815-835 kcal/day; approximately 43% carbohydrate, 29% protein, and 29% fat) formula diet product for 12 weeks, followed by a gradual food reintroduction phase combined with physical activity support for 12 weeks.
  Arms: Formula Diet
Other: Food-based diet — Participants will receive a low-calorie (815-835 kcal/day; 45-50% carbohydrate, 20-30% protein, and 20-30% fat) food-based diet created by dietitians for 12 weeks. After 12 weeks, participants will increase energy intake gradually and be encouraged to increase daily physical activity to maintain weight loss for another 12 weeks.
  Arms: Food-Based Diet

SUMMARY:
The prevalence of type 2 diabetes mellitus (T2DM) has been increasing rapidly in China. China currently has ~130 million diabetes cases, and over 90% are T2DM. T2DM is a leading cause of morbidity and mortality, posing substantial clinical and public health challenges. Reversing T2DM with a significant amount of weight loss via consuming a low-calorie diet is possible, but no studies have been conducted to determine whether low-calorie diets will help achieve significant weight loss and diabetes remission among Chinese patients with T2DM. The investigators design a pilot study to assess the feasibility of a low-calorie diet intervention program on weight loss and diabetes remission in a Chinese population with T2DM.

DETAILED DESCRIPTION:
Consistent evidence has shown that overweight and obesity are the leading cause of T2DM, which exacerbates the development of insulin resistance and disease progression. For overweight and obese patients with T2DM, there is a strong consensus that sustained and moderate weight loss can effectively improve glycemic control and blood pressure as well as reduce the need for glucose-lowering medications and improve quality of life.

Short-term dietary interventions using structured low-calorie diets (800-1,000 kcal/day) have shown to be an effective approach for losing weight and promoting sustained diabetes remission in T2DM patients who are overweight or obese. The United Kingdom DiRECT research team designed a structured, intensive intervention program of 12-20 weeks to achieve substantial weight loss and T2DM remission through energy restriction. Researchers recorded ≥15 kg of weight loss in 24% of the participants who underwent a low-calorie formula diet intervention (total diet replacement with 825-853 kcal/day formula low-energy diet meal replacement products). Among these participants, the diabetes remission rate reached 90%.

This non-randomized dietary intervention study comprises 2 study arms: a formula diet (815-835 kcal/day) and a food-based diet (815-835 kcal/day). Participants will be on either of the two low-calorie diets for 12 weeks to achieve at least 12 kg of weight loss (intensive weight loss phase). Participants may extend the weight loss phase if desired. After 12 weeks, participants in the formula diet group are allowed to consume actual meals gradually, and participants in both groups will increase their energy consumption gradually over the next 12 weeks (weight loss achievement and maintenance phase). Physical activity is recommended during the second phase for maintaining weight loss. This study is designed to assess feasibility of the low-calorie diet intervention, in preparation for a full-scale randomized control study. This pilot study also plans to explore potential mechanisms of the intervention for weight loss and diabetes remission.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed T2DM
* Most recent HbA1c level: 6.5%-12.0%
* Body mass index: 24-45 kg/m2
* Informed consent signed by participants in this study in accordance with requirements of local regulations and the Ethical Review Committee
* No plan to leave Shanghai in 2 years

Exclusion Criteria:

* Type 1 diabetes
* Current use of insulin and glucagon-like peptide-1 receptor agonists
* Major cardiovascular events (e.g., myocardial infarction, stroke, and heart failure) within the previous 6 months
* Weight loss >5 kg within the past 6 months
* Diagnosed eating disorders or any dieting behaviors
* Chronic kidney disease stage 3b or higher (estimated glomerular filtration rate <30 milliliter /min/1.73m2)
* Previously diagnosed psychiatric disorders, e.g., schizophrenia, post-traumatic stress disorder, obsessive-compulsive disorder, uncontrolled depression, uncontrolled epilepsy
* Severe arthritis and gout
* Gallstone disease or known asymptomatic gallstones
* Participation in another clinical research trial
* Being pregnant or have a positive pregnancy test result at screening, or have given birth within the past 90 days, or who are breastfeeding.
* Any known cancers
* Learning difficulties
* Alcoholism
* Pancreatitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Percent of adherence to the intervention | Baseline to 24 weeks
  Percent of adherence is calculated at the end of the intervention by dividing the number of participants who remain in and adhere to the intervention by the total number of participants who participate in the intervention.
Percent of participants achieving significant weight loss and diabetes remission | Baseline to 24 weeks
  Proportion of participants achieving significant weight loss (≥12kg) and diabetes remission, which is defined as having a glycated hemoglobin (HbA1c) level less than 6.5% while receiving no pharmacological therapy for diabetes for at least 3 months, will be estimated at 24 weeks.

SECONDARY OUTCOMES:
Aggregated safety assessment | Baseline to 24 weeks
  Glutathione, glutathione, total bilirubin, direct bilirubin, indirect bilirubin, urea nitrogen, creatinine, blood cell sorting count, urine routine, and adverse events are measured or recorded at the pre-specified time points to reflect number of participants with abnormal laboratory values and/or adverse events that are related to treatment.
Insulin sensitivity | Baseline to 24 weeks
  Insulin sensitivity is evaluated with insulin tolerance tests at the pre-specified time points.
Beta cell function | Baseline to 24 weeks
  Beta cell function is evaluated with arginine stimulation test at the pre-specified time points.
Level of fasting glucose | Baseline to 24 weeks
  Level of fasting glucose is measured using a blood sample from a finger stick when participants have an empty stomach (refraining from eating of drinking any liquids other than water for eight hours) at the pre-specified time points.
Level of postprandial glucose | Baseline to 24 weeks
  Level of postprandial glucose is measured using a blood sample from a finger stick two-hour later after participants eat their meals at the pre-specified time points.
Level of HbA1c | Baseline to 24 weeks
  Level of HbA1c is measured using a blood sample from a finger stick at the pre-specified time points.
Glucose homeostasis | Baseline to 24 weeks
  Time in Range, Time Above Range, and Time Below Range are measured at the pre-specified time points using continuous glucose monitor data.
Body fat composition and fat distribution | Baseline to 24 weeks
  Dual-energy X-ray absorptiometry scan is used for quantifying body composition. Magnetic resonance imaging scan is used to quantify fat in the liver and pancreas at the pre-specified time points.
Gut microbiota | Baseline to 24 weeks
  Metagenomic sequencing of fecal samples is performed to study gut microbiota including bacteria, fungi, archaea, and viruses at the pre-specified time points.
Traditional Chinese Medicine(TCM) tongue diagnosis estimated by tongue-face diagnosis instrument | Baseline to 24 weeks
  Parameters of tongue nature and tongue coating are estimated by tongue-face diagnosis instrument to detect hyperglycemic changes at the pre-specified time points.
TCM facial diagnosis estimated by tongue-face diagnosis instrument | Baseline to 24 weeks
  The changes of face complexion and surface gloss are estimated by tongue-face diagnosis instrument to reveal pathological changes of different viscera and bowels with different natures at the pre-specified time points.
Health-related quality of life | Baseline to 24 weeks
  The European Quality of Life 5-dimension 5-level questionnaire will be used to measure health-related quality of life at the pre-specified time points. The scale is numbered from 0 to 100. 100 measn the best health condition, and 0 means the worst health condition.
Diet | Baseline to 24 weeks
  The food frequency questionnaire will be used to assess diet and eating behaviors at the pre-specified time points.
Binge eating behaviors | Baseline to 24 weeks
  The binge eating scale will be used to assess the presence of binge eating behavior indicative of an eating disorder at the pre-specified time points (less than 17: non-binging; 18-26: moderate binging; 27 and greater: severe binging).
Diet and eating behaviors | Baseline to 24 weeks
  The three-factor eating questionnaire will be used to assess diet and eating behaviors at the pre-specified time points. All items are coded with either 0 or 1 point leading to maximum sum scores of 21 points for the domain of 'cognitive restraint', 16 points for 'disinhibition' and 14 points for 'hunger'. Higher scores indicate stronger characteristic values in the domains.
Psychological status-Anxiety | Baseline to 24 weeks
  The Self-Rating Anxiety Scale will be used to measure anxiety level at the pre-specified time points (20-44 normal range. 45-59 mild to moderate anxiety, 60-74 severe).
Psychological status-Depression | Baseline to 24 weeks
  Patient Health Questionaire-9 will be used to measure depression level at the pre-specified time points (0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe).
Sleep quality | Baseline to 24 weeks
  The Pittsburgh Sleep Quality Index will be used to measure sleep quality at the pre-specified time points. The scores range from 0 to 21 and a score >5 be considered as a significant sleep disturbance. Higher scores indicate worse sleep quality.
Metabolomic profiling performed by liquid chromatography mass spectrometry | Baseline to 24 weeks
  The liquid chromatography mass spectrometry (LC-MS) approach will be used to identify metabolites, pathways and networks that are associated with dietary interventions at the pre-specified time points. The major classes of metabolites including amino acids, carbohydrates, nucleotides, lipids, coenzymes, and cofactors are aggregated to demonstrate metabolic patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Wenze Zhong, Ph.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine; Feng Tao, Ph.D., Principal Investigator — Department of Endocrinology, Shanghai Municipal Hospital of Traditional Chinese Medicine
Locations (1):
- Department of Endocrinology, Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data materials will publish articles

REFERENCES:
- [Derived] Shi S, Wang S, Wu D, Li K, Yang G, Xu L, Feng N, Du X, Zhong VW. Epigenetic Signatures of Type 2 Diabetes Remission and Substantial Weight Loss: The Role of DNA Methylation in Response to Low-Calorie Diet Intervention. J Am Nutr Assoc. 2025 Nov-Dec;44(8):765-776. doi: 10.1080/27697061.2025.2513378. Epub 2025 Jun 5. PMID 40471649
- [Derived] Liu Z, Feng N, Wang S, Liu Y, Wang J, Tan Y, Dong Y, Sun Z, Du X, Xu Y, Tao F, Zhong VW. Low-calorie diets and remission of type 2 diabetes in Chinese: phenotypic changes and individual variability. Nutr J. 2025 Mar 14;24(1):42. doi: 10.1186/s12937-025-01101-z. PMID 40087696